CLINICAL TRIAL: NCT04525053
Title: Dosimetric Validation of Scans Generated by GAN From Pre-therapeutic MRI in Stereotactic Cerebral Radiotherapy (SBRT-IRM)
Brief Title: Dosimetric Validation of Scans Generated by GAN From Pre-therapeutic MRI in Stereotactic Cerebral Radiotherapy
Acronym: SBRT-IRM
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: SBRT-IRM ( 29BRC20.0156)
Record Dates: First submitted 2020-08-17; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stereotactic radiotherapy (SRT) is being widely accepted as a treatment of choice for patients with a small number of brain metastases and an acceptable size, allowing a better target dose conformity resulting in high local control rates and better sparing of organs at risk. Currently, imaging for such a delivery technique requires both a recent magnetic resonance imaging (MRI) brain study for volume definition and a computed tomography (CT) scan for SRT planning. An MRI-only workflow could reduce the risk of misalignment between the two imaging modalities and shorten the delay of planning. Given the absence of a calibrated electronic density on MRI, the investigators aim to assess the equivalence of synthetic CTs generated by a generative adversarial network (GAN) for planning in the brain SRT setting.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years old
* SRT treatment for one or more brain metastasis(ses)
* brain MRI and planning CT scans realized less than 14 days prior to the treatment delivery

Exclusion Criteria:

* MRI's field of view (FOV) judged insufficient for tumour(s) and OAR visualization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Restrospective inclusion of all patients treated with intra-cranial SRT for brain metastases from 2014 to 2018 in our single institution
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Local Gamma Analysis Passing Rate | Once, at the time of treatment delivery
  To be considered as comparable, 2 dose maps must have a Local Gamma Analysis Passing Rate higher than 98%. The primary outcome measure will be to compare the Local Gamma Analysis Passing Rate between the 2 dose maps (one initial dosimetric planification and one dosimetric planification extracted from the synthetic ct scan).

SECONDARY OUTCOMES:
Global Gamma Analysis Passing Rate | Once, at the time of treatment delivery
  To be considered as comparable, 2 dose maps must have a Global Gamma Analysis Passing Rate higher than 95%. The primary outcome measure will be to compare the Global Gamma Analysis Passing Rate between the 2 dose maps (one initial dosimetric planification and one dosimetric planification extracted from the synthetic ct scan).
Planning Target Volume's coverage values | Once, at the time of treatment delivery
  Planning Target Volume's (PTV) coverage values will be compared between the initial dosimetric planification and the dosimetric planification extracted from the synthetic ct scan.
Organs at risk Dose Constraints | Once, at the time of treatment delivery
  Dose constraints to the Organs at Risks (OAR) will be compared between the initial dosimetric planification and the dosimetric planification extracted from the synthetic ct scan.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 2 months and ending five years following the final study report completion.
Access Criteria: Data access request will be reviewed by the internal committee of Brest University Hospital. Requestor will be required to sign and complete a data access agreement.